CLINICAL TRIAL: NCT05400850
Title: The Effect of YOGA Asanas on Anterior and Posterior Myofascial Chain Activity in Elderly Individuals
Brief Title: YOGA Asanas and Myofascial Chain Activity in Elderly Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KaratatUH4
Record Dates: First submitted 2022-05-27; First posted 2022-06-02 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-05

CONDITIONS: Geriatrics
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YOGA (Experimental): sEMG values will record during different 5 YOGA Asana's
  Interventions: Other: YOGA

INTERVENTIONS:
Other: YOGA — Five different YOGA Asana's will made randomly

SUMMARY:
Aging is a differentiation process with chronological, biological, psychological and social characteristics, which occurs in the intrauterine period and ends with death. With aging, the structures and functions of tissues are affected and there is a decline in overall physical performance. Asanas in yoga use tonic muscle contraction coordinated with breath control and kinesthetic awareness, which saves energy compared to phasic muscle contraction often observed in physical exercises. We have not encountered a study examining the effect of asanas on muscular activity in old age. Our study will provide support to the literature in this direction.

DETAILED DESCRIPTION:
The study will be carried out on volunteers after the approval of the ethics committee. Before the research, individuals and / or their relatives will be informed about the purpose and content of the study. Participants will first start in mountain (Tadasana) asana. They will then be asked to come to the following asanas in a randomized order. In each of the asanas, you will statically pause for 15 seconds and repeat the movement three times. Participants will rest for 2 minutes between asanas. If deemed necessary during the application, modifications will be made in the movements and security measures will be taken. Warrior 2, elongated triangle, and Light Cluster stances will be evaluated for each limb separately. Muscle activations of individuals to the contralateral external oblique abdominal and ipsilateral adductor longus muscles of the anterior oblique myofascial chain lines and the contralateral latissimus dorsi and ipsilateral biceps femoris long head muscles to the posterior oblique myofascial chain lines will be evaluated using superficial EMG.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling male and female volunteers who do not do high-level exercise or take frequent long walks and do yoga

Exclusion Criteria:

* Active angina, uncontrolled hypertension, high resting heart rate or respiratory rate, unstable asthma, or exacerbated COPD; cervical spine instability or other significant neck injury, rheumatoid arthritis, unstable ankle, knee, hip, shoulder, elbow or wrist joints, hemiparesis or paraparesis, movement disorders (eg, Parkinson's disease), peripheral neuropathies, residual defective stroke, and severe vision or hearing problems, use of a walker or wheelchair, insufficient hearing to ensure safety in a yoga group setting

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
sEMG | During the YOGA Asana's
  sEMG activity will record during YOGA Asana's

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided